CLINICAL TRIAL: NCT04967092
Title: Efficacy and Safety of Modified Xiao-Feng Powder in the Treatment of Chronic Urticaria - A Double-Blind Randomized Placebo-Controlled Study
Brief Title: Modified Xiao-Feng Powder for Chronic Urticaria
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Lin Zhixiu (Other)
Responsible Party: Sponsor-Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C.Urticaria Study
Record Dates: First submitted 2021-07-14; First posted 2021-07-19 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Chronic Urticaria
Keywords: Chronic Urticaria; Chinese Medicines
MeSH Terms: conditions — Chronic Urticaria | interventions — Anti-Allergic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Xiao-Feng Powder (Active Comparator): Modified Xiao-Feng Powder granules will be taken twice daily for 12 weeks
  Interventions: Drug: Modified Xiao-Feng Powder + Antiallergics
- Placebo (Placebo Comparator): Placebo granules will be taken twice daily for 12 weeks
  Interventions: Other: Placebo + Antiallergics

INTERVENTIONS:
Drug: Modified Xiao-Feng Powder + Antiallergics — Modified Xiao-Feng Powder granules twice daily for 12 weeks plus Bilastine 20mg once daily for the first 6 weeks, and on-demand for the following 6 weeks.
  Arms: Modified Xiao-Feng Powder
Other: Placebo + Antiallergics — Placebo granules twice daily for 12 weeks plus Bilastine 20mg once daily for the first 6 weeks, and on-demand for the following 6 weeks.
  Arms: Placebo

SUMMARY:
Urticaria is a common skin disorder and 15-25% of people experience at least one attack of urticaria during their lifetime. Urticaria can be divided into acute urticaria (AU) and chronic urticaria (CU). CU is more common in adults, and affects women more frequently than men. According to Chinese medicine (CM) theory, CU is known as Yin Zhen. Nowadays, CM is widely used for managing CU in Hong Kong and mainland. Among different Chinese herbal formulae for urticaria, Xiao-Feng Powder (XFP), also known as Wind-Dispersing Powder, is one of the most frequently used Chinese herbal formulae for CU.

This study used modified Xiao-Feng Powder (mXFP) to evaluate the effectiveness and safety of mXFP in treating CU. Hence, a double-blind, randomised, placebo-controlled clinical trial design with strong scientific rigor will be employed in this study, and it would be able to provide robust clinical evidence on the efficacy and safety of mXFP for CU.

DETAILED DESCRIPTION:
Urticaria is a common skin disorder and 15-25% of people experience at least one attack of urticaria during their lifetime. Urticaria can be divided into acute urticaria (AU) and chronic urticaria (CU) according to the disease duration. CU is classified as either chronic autoimmune urticaria or chronic idiopathic urticaria.

In Chinese medicine theory, Urticaria is usually associated with either internal or external wind pathogen. Wind as a pathogenic factor is characterized by sudden onset and rapid changes in symptoms, and when resulting from an internal deficiency, it often leads to dryness.

Several research groups have conducted clinical studies to evaluate the efficacy of Chinese herbal medicine for the treatment of CU in recent decades. Among different Chinese herbal formulae for urticaria, Xiao-Feng Powder (XFP), also known as Wind-Dispersing Powder, is one of the most frequently used Chinese herbal formulae for CU, also has been widely used in Chinese medicine dermatology to expel wind and eliminate dampness, clear heat, nourish the blood and stop itchiness. Moreover, other researchers have found that XFP is effective in inhibiting inflammation, allergy, and oxidative stress in allergic skin diseases.

Investigators hypothesize that mXFP is effective and safe for the treatment of CU. In this study, eligible subjects will be randomized to receive either mXFP or placebo twice daily for 12 weeks followed by post-treatment visits at week 16. Subjects will take the standard therapy of antihistamines regularly for the first 6 weeks and then on on-demand basis for the next 6 weeks during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female;
2. Age from 18 to 65 years;
3. Documented history of CU for at least 6 weeks prior to entry in the study;
4. Meet EAACI/GA2LEN/EDF/WAO 2017 guidelines, i.e. spontaneous appearance of wheals, angioedema or both for > 6 weeks due to known or unknown causes;
5. Symptom severity must be greater than 10 points (UAS7 score);
6. Able to complete questionnaires and take medications as scheduled; and
7. Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Dual deficiency of Qi and blood according to Chinese medicine theory
2. Urticaria is induced by physical factors (e.g., cold urticaria, delayed pressure urticaria, solar urticaria, heat urticaria, vibratory angioedema) only;
3. Known to have dermatological diseases with skin pruritus;
4. Known to have any serious diseases such as cancer, severe kidney and liver impairments, autoimmune disease, thyroid disease, Hodgkin's disease, lymphoma, severe mental disorders, leukemia, and acute infectious disease;
5. Known to use oral/injectable corticosteroids, leukotriene inhibitors, immunosuppressants or other Chinese herbal medicine within one month of enrollment;
6. Known to receive omalizumab, ligelizumab, or other experimental biologic for CU;
7. Documented pregnancy or planning to conceive, breast-feeding women; or
8. Operate heavy machinery or need to drive motor vehicles as an essential part of their profession.
9. Know recent history (within previous 12 months) of drug addiction or alcohol abuse.
10. Involved in other interventional clinical studies at the same time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of Urticaria Activity Score (UAS7) | 12 weeks
  The UAS combines daily wheal numbers (0 = none, 1 = < 20 wheals/24 h, 2 = 20-50 wheals/24 h, and 3= > 50 wheals/24 h or large confluent areas of wheals), and pruritus intensity (0 = none, 1 = present but not annoying or troublesome, 2 = troublesome but does not interfere with normal daily activity or sleep, and 3 = severe pruritus, which is sufficiently troublesome to interfere with normal daily activity or sleep). The score ranges from 0 to 42 weekly. The highest score, the more severe of urticaria activity.

SECONDARY OUTCOMES:
Change of Urticaria Activity Score (UAS7) | 6 weeks and 16 weeks
  The UAS combines daily wheal numbers (0 = none, 1 = < 20 wheals/24 h, 2 = 20-50 wheals/24 h, and 3= > 50 wheals/24 h or large confluent areas of wheals), and pruritus intensity (0 = none, 1 = present but not annoying or troublesome, 2 = troublesome but does not interfere with normal daily activity or sleep, and 3 = severe pruritus, which is sufficiently troublesome to interfere with normal daily activity or sleep). The score ranges from 0 to 42 weekly. The highest score, the more severe of urticaria activity.
Change of Urticaria Control Test (UCT) | 6 weeks, 12 weeks and 16 weeks
  It collects retrospective information about the symptoms and quality of life impairment over the past 4 weeks. The lowest UCT score possible is 0 (no control) and the highest score possible is 16 (complete control). A score ≥12 indicates well-controlled urticaria, while a score of ≤11 points towards poor disease control.
Change of Visual Analog Scale of Itch Severity (VAS) | 6 weeks, 12 weeks and 16 weeks
  The VAS is a scale consisting of a 10 cm long line for measuring itch intensity and it has high reliability and concurrent validity. The highest score, the more itchiness.
Change of Urticaria Quality of Life Questionnaire (CU-Q2oL) | 6 weeks, 12 weeks and 16 weeks
  CU-Q2oL is a disease-specific questionnaire to measure the impact of disease on subjects' health-related quality of life in the last 2 weeks. The highest score, the poor quality of life.
Change of Angioedema Activity Score (AAS) | 6 weeks, 12 weeks and 16 weeks
  AAS is to assess disease activity in subjects with recurrent angioedema. The score ranges from 0 to 10 daily. The highest score, the more severe of the edema.
Change of Immunoglobulin E (IgE) test | 12 weeks
  To measure the change of IgE level between baseline and week 12
Change of microbiota test | 12 weeks
  To compare the presence and the relative amounts of some members of gut microbiota among patients with CU between baseline and week 12.
The use of concomitant drugs | Baseline, 6 weeks, 12 weeks and 16 weeks
  The dose of using the standard therapy of the antihistamines, Bilastine during study period will be compared between each study follow up visit throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine, The Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hung HY, Song T, Loo SKF, Chan KL, Ching JYL, Sum CH, Lo LCW, Chia SCP, Ho RTM, Cheong PK, Siu THC, Leung KC, Lin ZX. Efficacy and safety of modified Xiao-Feng Powder in the treatment of chronic urticaria: protocol of a randomized double-blind placebo-controlled study. Chin Med. 2022 Jul 22;17(1):87. doi: 10.1186/s13020-022-00642-3. PMID 35869554